CLINICAL TRIAL: NCT00003401
Title: Autologous Transplantation With Gemcitabine and High Dose BCNU Plus Melphalan Followed by Consolidation With DCEP Plus Gemcitabine and Taxol/Cisplatin in Patients With Multiple Myeloma and >12 Months of Standard Therapy
Brief Title: Peripheral Stem Cell Transplantation Plus Combination Chemotherapy in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: MSGCC-9731; CDR0000066405 (Registry Identifier: PDQ (Physician Data Query)); NCI-V98-1437
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Carmustine; Cisplatin; Cyclophosphamide; Dexamethasone; Etoposide; Gemcitabine; Melphalan; Paclitaxel; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: carmustine
Drug: cisplatin
Drug: cyclophosphamide
Drug: dexamethasone
Drug: etoposide
Drug: gemcitabine hydrochloride
Drug: melphalan
Drug: paclitaxel
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of peripheral stem cell transplantation plus combination chemotherapy in treating patients who have multiple myeloma that has been treated for longer than 12 months.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the complete and partial response in multiple myeloma patients receiving peripheral blood stem cells supported by gemcitabine and high dose carmustine and melphalan followed by consolidation therapy with gemcitabine plus cyclophosphamide/dexamethasone/etoposide/cisplatin (DCEP) and dexamethasone/paclitaxel/cisplatin. II. Evaluate the incidence of early death in comparison with historical data in this patient population. III. Evaluate the feasibility of chemotherapy with gemcitabine plus DCEP and dexamethasone/paclitaxel/cisplatin following autotransplantation in these patients.

OUTLINE: Patients receive gemcitabine IV over 100 minutes on day -5 and again 6 hours after administration of carmustine IV over 2 hours on day -2, followed by melphalan IV over 20 minutes on day -1. Patients receive intravenous CD34 peripheral blood stem cells on day 0. At 3 months and 9 months, patients with adequate hematologic counts receive cyclophosphamide IV, oral dexamethasone, etoposide IV, and cisplatin IV for 4 days. On day 3 of continuous infusions, gemcitabine is given over 100 minutes. At 6 and 12 months after autotransplant, patients receive oral dexamethasone on days 1-4, paclitaxel IV over 6 hours on day 2, and cisplatin IV over 24 hours on day 3. Patients are followed every 6 weeks to 3 months until death.

PROJECTED ACCRUAL: Approximately 24-63 patients will be accrued within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven multiple myeloma with greater than 12 months of prior therapy Bone marrow plasmacytosis at least 30% or protein criteria present No obvious myelodysplastic changes in the bone marrow No CNS disease

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: SWOG 0-2 (3-4 acceptable if based solely on bone pain) Life expectancy: Not specified Hematopoietic: CD34+ at least 4,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT or SGPT no greater than 4 times upper limit of normal No active or chronic hepatitis or liver cirrhosis Renal: Creatinine no greater than 3.0 mg/dL Cardiovascular: LVEF greater than 50% Pulmonary: FEV1 or FVC at least 50% of predicted DLCO at least 50% of predicted Patients unable to complete pulmonary function tests must have a CT scan of the chest and acceptable arterial blood gases of PO2 greater than 70 Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception HIV negative No active infection requiring IV antibiotics

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy Endocrine therapy: Prior steroid therapy allowed Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01 (Actual); Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry R. Meisenberg, MD, Study Chair — University of Maryland Greenebaum Cancer Center
Locations (1):
- Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland, United States